CLINICAL TRIAL: NCT00960362
Title: A Randomised, Double-blind, Placebo-controlled, and Single Dose-escalation Trial of AGS-009 Administered in Subjects With Systemic Lupus Erythematosus
Brief Title: An Investigation of AGS-009 in Patients With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Argos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AGS-009-001
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Inflammation; Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Inflammation; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- A (Placebo Comparator)
  Interventions: Drug: placebo
- B (Experimental): Intravenous cohort 1; 0.01 mg/kg
  Interventions: Drug: AGS-009
- C (Experimental): Intravenous cohort 2; 0.1 mg/kg
  Interventions: Drug: AGS-009
- D (Experimental): Intravenous cohort 3; 0.6 mg/kg
  Interventions: Drug: AGS-009
- E (Experimental): Intravenous cohort 4; 3.0 mg/kg
  Interventions: Drug: AGS-009
- F (Experimental): Intravenous cohort 5; 10 mg/kg
  Interventions: Drug: AGS-009
- G (Experimental): Intravenous cohort 6; 30 mg/kg
  Interventions: Drug: AGS-009

INTERVENTIONS:
Drug: AGS-009 — Single dose in the range of 0.01 to 30 mg/kg administered intravenously (in the vein)
  Arms: B; C; D; E; F; G
Drug: placebo — Single dose of 0 mg/kg administered intravenously (in the vein) cohort 1-6.
  Arms: A

SUMMARY:
This trial is conducted in North America. The aim of this clinical trial is to investigate the safety, tolerability, pharmacokinetic and signs of bioactivity of increasing single doses of AGS-009 in patients with systemic lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE
* Disease duration longer or equal to 6 months
* Stable, mild to moderate active SLE
* Receiving stable maintenance therapy

Exclusion Criteria:

* Significant lupus nephritis
* Active central nervous system (CNS) disease
* Significant arterial or venous thrombosis (blood clots) within 12 months prior to dosing
* Active vasculitis requiring treatment
* Body weight over 120 kg
* History of cancer
* Infections
* viral: HIV, hepatitis B or C, Epstein-Barr virus (EBV), cytomegalovirus (CMV), varicella zoster virus (VZV), or herpes simplex virus (HSV-1 or HSV-2)
* tuberculosis (TB)
* Severe systemic microbial infections within the past 12 months prior to dosing
* Immunosuppressive and immune modulating therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | From dosing at visit 2 until end of safety visits at visit 8.

SECONDARY OUTCOMES:
Pharmacokinetic - AUC (area under the curve) | From dosing at visit 2 until end of safety visits at visit 8.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Miesowicz, Ph.D., Study Director — Argos Therapeutics
Locations (6):
- United States (6):
  - Birmingham, Alabama
  - Kansas City, Kansas
  - Lake Success, New York
  - Durham, North Carolina
  - Duncansville, Pennsylvania
  - Dallas, Texas

REFERENCES:
- See also: Argos Therapeutics — http://www.argostherapeutics.com